CLINICAL TRIAL: NCT03039608
Title: Effect of a Combination of Local Steroid Injection With Oral Steroid Administration for the Prevention on Esophageal Stricture After Endoscopic Submucosal Dissection for Early Esophageal Neoplasm：a Randomized Controlled Trial
Brief Title: Effect of a Combination of Local Steroid Injection With Oral Steroid Administration for the Prevention on Esophageal Stricture After Endoscopic Submucosal Dissection for Early Esophageal Neoplasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: xmdrct
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Esophageal Stricture
Keywords: esophageal stricture; endoscopic submucosal dissection; prevention
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination group (Experimental): combination of local steroid injection（triamcinolone ）with oral steroid administration（prednisone）
  Interventions: Drug: combination of local steroid injection（triamcinolone ）with oral steroid administration（prednisone）
- control group (Active Comparator): oral steroid administration（prednisone）
  Interventions: Drug: oral steroid administration（prednisone）

INTERVENTIONS:
Drug: combination of local steroid injection（triamcinolone ）with oral steroid administration（prednisone） — local steroid injection and oral steroid
  Arms: combination group
Drug: oral steroid administration（prednisone） — oral steroid
  Arms: control group

SUMMARY:
The method of esophageal endoscopic submucosal dissection (ESD) to remove superficial esophageal neoplasms has gained widespread acceptance as an alternative to surgery recently these years especially in Asian countries. However, besides of perforation and bleeding, another complication postoperative esophageal stricture is frequently observed after the removal of large-sized esophageal neoplasms by ESD. Dysphagia caused by postoperative stricture substantially decreases the patient's quality of life, requiring further therapy. Although the exact incidence is unknown, esophageal stricture is supposed to be related to the extent of the circumference being resected. In previous study by Ono et al，it is reported that 90% of patients with lesions of circumferential extension of more than three-fourths experienced postoperative stricture after esophageal ESD. There were some reported studies exploring new ways to prevent esophageal stricture after ESD, such as oral prednisolone and local corticosteroid injection. Corticosteroids can inhibit not only collagen synthesis but also enhance collagen breakdown, thereby inhibiting stricture formation. Some studies reveled that just oral prednisolone oral is effective option for the prevention of post-ESD stricture. However, most of the reported studies were non RCTs with small sample. In the primary study, the investigators search a new method of combination of both oral and local injection to prevent esophageal stricture，as a result，stricture at 8 weeks after ESD was found in 19 of 36 patients in the no corticosteroid group but only 4 of 34 in the corticosteroid group. Unfortunately，the study was also retrospective. So, the investigators plan to undertake a prospective, randomized controlled trial to evaluate the prophylactic effects of combination of local steroid injection with oral steroid administration for esophageal stenoses complicating extensive ESD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who has undergone esophageal ESD
2. Histologically confirmed early squamous cell carcinoma or high grade intraepithelial neoplasia of the esophagus
3. ESD resulted in a mucosal defect involving more than two-thirds of the esophageal circumference.

Exclusion Criteria:

1. Severe circulatory or respiratory disease，severe renal impairment
2. Women in pregnancy and lactation
3. Patients with steroid contraindications
4. Patients refuse to join in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
the stricture rate | 12weeks
  the incidence of esophageal rate after ESD
the time when stricture occurs | 12weeks

SECONDARY OUTCOMES:
the frequency of dilatation sessions required | 12 months
  the frequency of dilatation sessions required after stricture
the frequency of complications | 12 months
  complications related with steroid administrations or the process of ESD

CONTACTS AND LOCATIONS:
Overall Officials: Meidong Xu, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China